CLINICAL TRIAL: NCT05834452
Title: Treatment of Posterior Benign Paroxysmal Positional Vertigo With Mechanical Rotational Chair: A Randomized Controlled Trial Comparing Epley and 360° Maneuvers.
Brief Title: Treatment of Posterior Benign Paroxysmal Positional Vertigo With Mechanical Rotational Chair.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Malene Hentze Hansen, medical doctor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220060
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Benign Paroxysmal Positional Vertigo; BPPV
Keywords: Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular Diseases; Epley Maneuver; TRV chair; Mechanical Rotational Chair
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Epley Maneuver (Active Comparator): Treatment of BPPV with the Epley Maneuver in the TRV chair. No kinetic energy will be used.
  Interventions: Procedure: The Epley Maneuver; Device: Mechanical rotational chair
- the 360 Maneuver (Active Comparator): Treatment of BPPV with the 360 Maneuver in the TRV chair.
  Interventions: Procedure: The 360 Degree Maneuver; Device: Mechanical rotational chair

INTERVENTIONS:
Procedure: The Epley Maneuver — 5 step procedure where the patient:
  1. Sits upright in a neutral position
  2. Rotate 45° towards the affected side around the yaw axis and then ro-tate 135° backward around the pitch axis
  3. Rotated 90° towards the unaffected side around the yaw axis
  4. Rotate a further 90° toward the unaffected side around the yaw axis
  5. Rotates back to an upright position with a 135° backward rotation around the pitch axis.
  Arms: the Epley Maneuver
Procedure: The 360 Degree Maneuver — 5 step procedure where the patient:
  1. Sits upright in a neutral position
  2. Rotate 45° towards the affected side around the yaw axis and then ro-tate 135° backward around the pitch axis
  3. Rotate a further 90° backward around the pitch axis (total 225°)
  4. Rotate a further 90° backward around the pitch axis (total 315°)
  5. Rotate back to an upright position with an additional 45° backward rota-tion around the pitch axis (total 360°).
  Arms: the 360 Maneuver
Device: Mechanical rotational chair — TRV chair

SUMMARY:
Comparison of treatment efficacy of Epley maneuver and 360 maneuver in a mechanical rotational chair (TRV chair) in patient with posterior benign paroxysmal positional vertigo (BPPV).

DETAILED DESCRIPTION:
Open-label, randomized controlled trial comparing the Epley maneuver with the 360 maneuver using the TRV chair in both scenarios. Patients diagnosed with posterior BPPV will be randomized to receive treatment with either the Epley maneuver or the 360 maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Confirmed unilateral p-BPPV (canalithiasis and cupulolithiasis)
* Understand written and spoken Danish

Exclusion Criteria:

* Pregnancy
* Weight ≥ 150 kg and or Height ≥ 2m
* Not possible to attend follow-up visits
* Insufficient cooperation during diagnostic testing or treatment in the mechanical rotational chair
* Have received treatment for BPPV in a mechanical rotational chair within the last 6 months
* Sedative antihistamines are taken within the past 7 days
* Comorbidities: Heart failure (EF<40), known cerebral aneurysm, cerebrovascular events (<3 months), and dissection disease
* Spontaneous or gaze evoked nystagmus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment success after first treatment | 2 year
  Number of subjects achieving resolution of vertigo and nystagmus after one treatment
Number of treatments | 2 year
  Number of treatment necessary to achieve resolution of vertigo and nystagmus

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) Questionnaire | 2 year
  Comparison of pre-treatment score and post-treatment score
Adverse events | 2 year
  Registration of adverse events
Recurrence rate | 2 year
  Recurrence of BPPV 3 and 6 months after successful treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Malene Hentze Hansen, MD, Principal Investigator — Department of Otolaryngology, Head & Neck Surgery and Audiology
Locations (1):
- epartment of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No